CLINICAL TRIAL: NCT06807671
Title: Does Planned Visual Training Affect the Attitudes, Beliefs and Symptoms of Individuals with Heart Failure Towards Their Disease?
Brief Title: Effect of Planned Visual Training on Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Dilan Deniz Akan, PhD, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCBU dilan deniz akan
Record Dates: First submitted 2024-12-26; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
Keywords: heart failure; health belief model; patient training; nursing
MeSH Terms: conditions — Heart Failure | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the study do not know whether they are in the experimental or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): No Intervention: Control group No intervention was made by the researcher during the study. Only data was collected. At the end of the study, visual training based on the planned Health Belief Model was given and all patients who continued the study were given brochures and heart-shaped key chains designed by the researchers.
- Experimental Group (Experimental): Experimental: intervention group The sample of this simple-randomized controlled experimental study consisted of heart failure patients who applied to Manisa Celal Bayar University (MCBU) Hafsa Sultan Hospital Cardiology Polyclinic between September 2021 and March 2022. Patients who were determined by drawing lots according to their protocol numbers using the simple random sampling method were assigned to the intervention group. Patients assigned to the intervention group were given planned training based on the Health Belief Model. The intervention group was followed up for six months. A total of three interviews were conducted with the intervention group (First interview, 3rd month interview and 6th month interview).
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — Patients in the intervention group received HBM based training for a period of 6 months. During the training, one-on-one interviews were provided with each patient. Patients were shown a power point presentation, a brochure, and 3 training videos. Any questions patients had were answered one-on-one.
  Other Names: Educational intervention
  Arms: Experimental Group

SUMMARY:
This study was conducted to evaluate the effects of planned visual education based on the Health Belief Model on the attitudes, beliefs, and symptoms of heart failure patients towards their disease. Planned visual education based on the Health Belief Model has positive effects on the attitudes, beliefs, and symptoms of heart failure patients towards their disease.

DETAILED DESCRIPTION:
This study, which evaluated the effects of planned visual education based on the Health Belief Model on the attitudes, beliefs, and symptoms of patients with heart failure towards their disease, was conducted with 110 heart failure patients. The study was planned as a randomized controlled experimental study conducted on two groups as intervention (n = 55) and control group (n = 55). The study was conducted between September 2021 and March 2022 at Manisa Celal Bayar University (MCBU) Hafsa Sultan Hospital Cardiology Polyclinic. Simple randomization method was used in assigning the sample group to the experimental and control groups. Data were collected using "the Patient Identification Form", "the Health Belief Model Scale - Heart Failure" and "Memorial Symptom Assessment Scale - Heart Failure".

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65,
* Those with no communication problems,
* Those diagnosed with NYHA I-II heart failure,
* Those without cognitive impairment,
* Those who can understand and speak Turkish,
* Those who agree to participate in the study.

Exclusion Criteria:

* Patients who do not agree to participate in the study,
* Patients who want to leave the study,
* Patients with NYHA III-IV heart failure diagnosis,
* Patients diagnosed with cancer,
* Patients with diabetic foot or amputation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Data collection tool | Pre-test
  In order to monitor the effectiveness of the intervention in the study, a 6-month follow-up was conducted and data were collected from the intervention group 3 times (before the intervention, at 3 months and at 6 months) and from the control group twice (at the first interview and at 6 months) through data collection forms.
  HBM-based education program was applied to the intervention group as an intervention.
  Data collection tools were "Patient Information Form", "Memorial Symptom Assessment Scale - Heart Failure (MSAS-HF)" and "Health Belief Model Scale in Heart Failure (HBM-HF)".
  Patient Information Form: A total of 15 questions are included, including sociodemographic information (such as age, gender, marital status, education status, employment status, occupation and income status) and additional information regarding HF/HF treatment (perceived health status, compliance with diet, exercise, treatment compliance, regular doctor visits, etc.) of the participants.

SECONDARY OUTCOMES:
Data collection tool | 3 month
  In the study, 3-month data were collected from the intervention group using the same measurement tools.
  MSAS-HF: The scale is used to evaluate the symptoms experienced by patients with HF. It consists of three sub-dimensions in total (physical symptoms, psychological symptoms, and HF symptoms). For the symptoms encountered, it is expected to rate the frequency and severity of the symptom with a four-point Likert-type assessment, and the discomfort with a five-point Likert-type assessment. In the calculation, symptom load is first calculated for each symptom. The load of the unseen symptom is evaluated as zero. The Cronbach alpha values of the scale were reported as 0.53 for physical symptoms, 0.63 for psychological symptoms, and 0.55 for HF symptoms.

OTHER OUTCOMES:
Data collection tool | 6-months / Post-test
  In the 6th month of the study, after the educational intervention was completed, data were collected again from the intervention and control groups through data collection forms.
  HBM-HF: The scale was developed to assess the attitudes and beliefs of HF patients towards their disease. The scale consists of 24 items and five sub-dimensions (perceived susceptibility, perceived severity, perceived benefits, perceived barriers, self-efficacy) and is a five-point Likert-type scale. The items of the perceived barrier sub-dimension in the scale are reverse coded. The scale does not have a total score and each sub-dimension is calculated independently. Higher scores indicate higher perception of susceptibility, perceived severity, perceived benefits, and good self-efficacy, while lower scores indicate stronger perception of barriers. The Cronbach's alpha coefficients of the sub-dimensions are 0.91, 0.86, 0.88, 0.75, and 0.84, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It can be shared upon request, if the relevant ethics committee approves.
Supporting Information: CSR
Time Frame: starting 6 months after publication
Access Criteria: It can be shared upon request, if the relevant ethics committee approves.